CLINICAL TRIAL: NCT03466359
Title: Nutritional Responses to Chronic Exercise- Versus Energy Restriction-induced Energy Deficits in Obese Adolescents
Brief Title: Energy Intake and Energy Deficit in Obese Adolescents
Acronym: IDEFIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Tza Nou - Maison médicale pour enfants et adolescentes - 230, rue Vercingétorix - B.P. 77 - 63150 La Bourboule (Unknown); SSR Nutrition-Obésité - 33-35 rue Maréchal Leclerc - 63000 Clermont-Ferrand (Unknown); Laboratoire AME2P. Campus universitaire des cezeaux, 63170 Aubiere, Cedex (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-378; 2017-A00817-46 (Other: 2017-A00817-46)
Record Dates: First submitted 2018-02-08; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Pediatric Obesity
Keywords: appetite control; obesity; Adolescents; Physical activity
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEF-EI (Experimental): these adolescents will follow a dietary restriction of 10% of their daily energy intake.
  Interventions: Behavioral: DEF-EI : Energy restriction induced energy deficit
- DEF-EX (Experimental): these adolescents will increase their physical activity-induced energy expenditure by 10% per day.
  Interventions: Behavioral: DEF-EX : Exercise induced energy deficit

INTERVENTIONS:
Behavioral: DEF-EI : Energy restriction induced energy deficit — DEF-EI : Energy restriction induced energy deficit The content of their energy intake will be decreased by 10% daily compared with the phase one of the protocol (stabilization of intake). This decrease will be allowed by the internship nature of the clinical program; all the meals are prepared and served by the personal of the clinical centre.
  Arms: DEF-EI
Behavioral: DEF-EX : Exercise induced energy deficit — DEF-EX : Exercise induced energy deficit While their intake will remain the same as phase 1, they will increase their physical activity energy expenditure by 10% thanks to an increase of their prescribed exercise intensities or durations.
  Arms: DEF-EX

SUMMARY:
The aim of the present study is to compare the effect of two weight loss interventions inducing the same energy deficit but one based on exercise and one using dietary restriction, on appetite control in obese adolescents. Investigator hypothesis that daily energy intake and hunger will be increased in the dietary restriction group but not in response to the exercise program.

DETAILED DESCRIPTION:
The present study will compare the nutritional responses to two 4-month weight loss programs inducing the same energy deficit in obese adolescents, one based on exercise and the other one using dietary restriction. After a first 4-month phase stabilizing the adolescents' daily energy intake and expenditure, half of the sample with increase their physical activity to induce a 10% increase of their daily energy expenditure (maintaining the same energy intake) while the other half will stick with the same physical activity program but reduce their daily intake to match for the same 10% energy deficit. Before, at the end and 4 months after the intervention, Investigator will assess the adolescents' energy intake and appetite control by measuring: ad libitum energy intake, appetite feelings throughout the day, food preferences, food reward. But also all the potential underneath mechanisms based on gastro-peptides and adipokines. Finally, sleep metabolism will be assessed using polysomnography as a potential link between weight loss and appetite control. Body composition, quality of life, aerobic capacities and resting metabolic rate will also be measured at each time point.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in energy intake at lunch time | Before, after 10 months and 4 month after the intervention
  food intake will be measured ad libitum during a lunch time buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be assessed by a member of the investigation team

SECONDARY OUTCOMES:
change in FM | Before, after 10 months and 4 month after the intervention
  Fat mass (FM) was assessed using DXA following standardized procedures
Aerobic capacity | Before, after 10 months and 4 month after the intervention
  VO2peak will be measured during a graded exhaustive cycling test performed by a specialized medical investigator from the Department of Sports Medicine, Functional and Respiratory Rehabilitation (Clermont-Ferrand University Hospital). The initial power will be set at 30 W for three minutes and followed by 15 W increments every 1.5 minutes.
Insulin concentration | Before, after 10 months and 4 month after the intervention
  : Insulin will be assessed thanks to a fasting blood sample taken by a specialized nurse.
Glycaemia concentration | Before, after 10 months and 4 month after the intervention
  glycaemia, will be assessed thanks to a fasting blood sample taken by a specialized nurse.
total cholesterol concentration | Before, after 10 months and 4 month after the intervention.
  cholesterol total will be assessed thanks to a fasting blood sample taken by a specialized nurse.
HDL-C concentration | Before, after 10 months and 4 month after the intervention
  HDL-C will be assessed thanks to a fasting blood sample taken by a specialized nurse
LDL-C concentration | Before, after 10 months and 4 month after the intervention
  LDL-C will be assessed thanks to a fasting blood sample taken by a specialized nurse.
Triglycerides concentration | Before, after 10 months and 4 month after the intervention
  Triglycerides concentration will be assessed thanks to a fasting blood sample taken by a specialized nurse.
Acylated Ghrelin concentration | Before, after 10 months and 4 month after the intervention
  Acylated Ghrelin concentration will be assessed thanks to a fasting blood sample taken by a specialized nurse
Leptin concentration | Before, after 10 months and 4 month after the intervention
  Leptin concentration will be assessed thanks to a fasting blood sample taken by a specialized nurse
Sleep metabolism | Before, after 10 months and 4 month after the intervention
  sleep duration will be assessed during an overnight polysomnography.
appetite feelings | Before, after 10 months and 4 month after the intervention
  hunger satiety will be assessed using visual analogue scale at regular interval through a test day
Quality of life Score | Before, after 10 months and 4 month after the intervention
  A total Quality of life score will be obtain thanks to the "SF36" questionnaire. This is a self-reported questionnaire. A member of the investigation team will be present to help and guide the adolescents if needed
Health Perception | Before, after 10 months and 4 month after the intervention
  A total Health Perception score will be obtain thanks to the "Health Perception Questionnaire ". This is a self-reported questionnaire. A member of the investigation team will be present to help and guide the adolescents if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Roche J, Corgosinho FC, Damaso AR, Isacco L, Miguet M, Fillon A, Guyon A, Moreira GA, Pradella-Hallinan M, Tufik S, Tulio de Mello M, Gillet V, Pereira B, Duclos M, Boirie Y, Masurier J, Franco P, Thivel D, Mougin F. Sleep-disordered breathing in adolescents with obesity: When does it start to affect cardiometabolic health? Nutr Metab Cardiovasc Dis. 2020 Apr 12;30(4):683-693. doi: 10.1016/j.numecd.2019.12.003. Epub 2019 Dec 16. PMID 32008915